CLINICAL TRIAL: NCT07197242
Title: Assessment of Lipoprotein(a) in Patients Undergoing Elective Percutaneous Coronary Revascularization: Implications for Cardiovascular Risk Stratification
Brief Title: Prognostic Role of Lipoprotein(a) in Elective Percutaneous Coronary Revascularization
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ahmed gamal abdelhakeem ahmed, resident at Cardiology Department, Assiut University
Other Study IDs: Lp(a) and Risk in Elective PCI
Record Dates: First submitted 2025-09-20; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: PCI
Keywords: PCI; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients (≥18 years old) undergoing elective PCI for stable coronary artery disease will form: The targeted cohort consists of men and women presenting with stable ischemic heart disease scheduled to undergo elective PCI at the Assiut University Heart Hospital cardiac catheterization unit

SUMMARY:
The study investigates the role of Lipoprotein(a) [Lp(a)] levels in predicting cardiovascular risk and adverse events in patients undergoing elective percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
his is a multicenter prospective observational cohort study conducted at Assiut University Heart Hospital and affiliated centers. The study focuses on patients undergoing elective (non-ACS) PCI for stable coronary artery disease. Baseline Lp(a) levels will be measured pre-PCI using isoform-insensitive immunoassays, and patients will be followed for 24 months to document cardiovascular outcomes. The primary goal is to assess whether elevated Lp(a) (≥125 nmol/L) independently predicts 2-year major adverse cardiovascular events (MACE) beyond conventional risk factors and procedural complexity. The study also aims to evaluate the prevalence of elevated Lp(a) among this population and its incremental prognostic value for refining risk stratification models such as SYNTAX II/ACEF. Collected blood samples will be stored in a biobank for future exploratory analyses.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older

Undergoing elective PCI for stable coronary artery disease

Ability to provide informed consent

Willingness to undergo blood sampling prior to PCI

Exclusion Criteria:

* Acute coronary syndrome within 30 days

Cardiogenic shock

Prior heart transplant or left ventricular assist device (LVAD)

Life expectancy less than 1 year due to non-cardiac causes

Participation in a blinded Lp(a)-lowering outcome trial at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: targeted cohort consists of men and women presenting with stable ischemic heart disease scheduled to undergo elective PCI at the Assiut University Heart Hospital cardiac catheterization unit. Eligible patients must provide informed consent and undergo baseline blood sampling. The study excludes patients with recent acute coronary syndrome (ACS within 30 days), cardiogenic shock, prior cardiac transplantation/LVAD, limited life expectancy from non-cardiac causes, or those enrolled in contemporary blinded clinical trials specifically for Lp(a)-lowering therapies. By selecting an elective CAD population, the study narrows focus to a lower baseline
Sampling Method: Probability Sample
Enrollment: 156 (Estimated)
Dates: Start 2026-10-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of major adverse cardiovascular events (MACE) | one year
  Incidence of all non-fatal myocardial infarction, and ischemia-driven target vessel revascularization or or definite/probable stent thrombosis.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vinci P, Di Girolamo FG, Panizon E, Tosoni LM, Cerrato C, Pellicori F, Altamura N, Pirulli A, Zaccari M, Biasinutto C, Roni C, Fiotti N, Schincariol P, Mangogna A, Biolo G. Lipoprotein(a) as a Risk Factor for Cardiovascular Diseases: Pathophysiology and Treatment Perspectives. Int J Environ Res Public Health. 2023 Sep 6;20(18):6721. doi: 10.3390/ijerph20186721. PMID 37754581